CLINICAL TRIAL: NCT02969811
Title: Cardiac Injury and Anaemia Following Surgery for Fractured Neck of Femur: An Observational Study Study Protocol: Cardiac Injury and Anaemia Following Surgery for Fractured Neck of Femur: An Observational Study
Brief Title: Cardiac Injury and Anaemia Following Surgery for Fractured Neck of Femur: An Observational Study Study Protocol: Cardiac Injury and Anaemia Following Surgery for Fractured Neck of Femur
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC16087
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Last update posted 2024-09-24 (Actual); Status verified 2016-11

CONDITIONS: Anaemia, Myocardial Ischaemia, Fractured Neck of Femur
MeSH Terms: conditions — Anemia; Coronary Artery Disease; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Severely Anaemic: Patients with Hb 90 g/L or less
- Non-Anaemic: Patients with Hb greater than 90 g/L

SUMMARY:
Blood transfusion is an expensive and finite resource and optimum transfusion threshold in surgical patients is yet to be defined. Patients commonly receive blood transfusions to reduce the risk of myocardial ischaemia or improve perfusion of other organs (e.g. the kidneys), but this treatment may have important adverse effects including postoperative infection. Patients undergoing surgery for fractured neck of femur are often elderly, with co-morbidities and a high risk of postoperative complications, including MI and AKI. We propose to conduct a study with the following aims:

1. To describe the incidence of anaemia and transfusion in patients undergoing surgery for fractured neck of femur.
2. To use clinical and biochemical data to measure the incidence of perioperative cardiac and kidney injury in this group.
3. To evaluate highly sensitive serum troponin and urinary MALDI-MS as possible endpoints in a future prospective randomised trial of perioperative transfusion.

DETAILED DESCRIPTION:
Blood transfusion is an expensive and finite resource and optimum transfusion threshold in surgical patients is yet to be defined. Patients commonly receive blood transfusions to reduce the risk of myocardial ischaemia or improve perfusion of other organs (e.g. the kidneys), but this treatment may have important adverse effects including postoperative infection. There is great interest in restrictive transfusion practices (e.g. a transfusion trigger of 70 g L-1), however patients with co-existing cardiovascular disease have been excluded from studies of restrictive versus liberal transfusion strategies. Highly sensitive troponin assays are now available, which allow clinicians to reliably detect cardiac injury in increased numbers of patients who have undergone major surgery. Troponin release after surgery is common, as high as 40% in some studies. Patients undergoing surgery for fractured neck of femur are often elderly, with co-morbidities and a high risk of postoperative complications, including MI and AKI. We propose to conduct a study with the following aims:

1. To describe the incidence of anaemia and transfusion in patients undergoing surgery for fractured neck of femur.
2. To use clinical and biochemical data to measure the incidence of perioperative cardiac and kidney injury in this group.
3. To evaluate highly sensitive serum troponin and urinary MALDI-MS as possible endpoints in a future prospective randomised trial of perioperative transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Fractured Neck of Femur
* Age >50
* Informed consent

Exclusion Criteria:

* refusal of consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered fractured neck of femur.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Cardiac Injury | 72 hours after surgery
  Serum Troponin above upper reference limit

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT02969811/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT02969811/ICF_001.pdf